CLINICAL TRIAL: NCT03735147
Title: Assessment of Viral Shedding Week Following Administration of Live Attenuated Influenza Vaccine in Children: FluSHED-2 Study
Brief Title: Assessment of Viral Shedding Week Following Administration of Live Attenuated Influenza Vaccine in Children
Acronym: FluSHED-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18SM4658; 2018-002470-42 (EudraCT Number); 18/LO/1317 (Other: NHS HRA)
Record Dates: First submitted 2018-10-22; First posted 2018-11-08 (Actual); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Influenza Vaccines
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All children (Experimental): Administration of live attenuated influenza vaccine (LAIV)
  Interventions: Biological: Live attenuated influenza vaccine (LAIV)

INTERVENTIONS:
Biological: Live attenuated influenza vaccine (LAIV) — Single dose of LAIV
  Other Names: Fluenz Tetra

SUMMARY:
LAIV shedding studies in children could be an important way to confirm whether impediments to viral replication do indeed explain these observed reductions in vaccine effectiveness (VE), whether prior vaccination has any influence on replication and what future implications (if any) this might have for the UK paediatric LAIV programme. LAIV virus replication in children will be dependent on virological and host factors. The virus factors include replicative fitness of individual strains and the susceptibility to inhibition by other replicating strains (ability to compete). Host factors which may influence this include pre-existing specific immunity as a result of prior infection or previous vaccination (with either LAIV or IIV), and innate immune factors including mucosal immunity.

There is significant variability in shedding across viral subtypes in studies done to date, so there is a need to obtain local data in a small pilot observational study which will look in detail at virus shedding by sequential daily virus samples, something not possible on a larger scale. The data generated will inform future LAIV studies in the UK in terms of optimum time of sample collection for viral shedding studies, which are likely to be required on a regular basis, to supplement field studies of vaccine effectiveness.

This study will enrol up to 30 children that will allow these factors to be assessed. Both written informed consent from parent/ guardian and written assent from the child will be in place prior to any study procedure. All participants will have a baseline assessment of pre--existing influenza immunity (blood test, oral fluid collection and nasal swabs), followed by a single dose of LAIV. Parents will then be asked to take nasal swabs at home on days 1, 2, 3, 4, 5, 6, 7, 8, with further nasal swab, blood test and oral fluid collection in hospital 4 weeks later, in order to assess for immune responses to LAIV.

ELIGIBILITY:
Inclusion Criteria:

* Children age 6 years to 15 years +364 days of age on enrolment
* Children eligible to receive LAIV in accordance with current UK vaccine policy
* Written informed consent given by parent/ guardian and assent from child

Exclusion Criteria:

Contraindications to LAIV (notwithstanding allergy to egg protein), which include:

* Hypersensitivity to the active ingredients, gelatin or gentamicin (a possible trace residue)
* Previous systemic allergic reaction to LAIV
* Previous allergic reaction to an influenza vaccine (not LAIV) is a relative contra-indication, which must be discussed with the CI to confirm patient suitability
* Children/adolescents who are clinically immunodeficient due to conditions or immunosuppressive therapy such as: acute and chronic leukaemias; lymphoma; symptomatic HIV infection; cellular immune deficiencies; and high-dose corticosteroids*.
* Children / adolescents younger than 18 years of age receiving salicylate therapy because of the association of Reye's syndrome with salicylates and wild-type influenza infection.
* Pregnancy (determined by history). Where this cannot be confirmed, a urine pregnancy test will be performed.

  * High---dose steroids is defined as a treatment course for at least one month, equivalent to a dose greater than 20mg prednisolone per day (any age), or for children under 20kg, a dose greater than 1mg/kg/day.

NB: LAIV is not contraindicated for use in individuals with asymptomatic HIV infection; or individuals who are receiving topical/inhaled/low-dose oral systemic corticosteroids or those receiving corticosteroids as replacement therapy, e.g. for adrenal insufficiency.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Turner, FRACP, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust (St. Mary's Hospital), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Children
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Children
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — LAIV vaccination in previous years
  Participants
    United Kingdom | 12

OUTCOME MEASURES:

1. Primary Outcome: Type-specific Vaccine Virus Shedding in 2018/19 - Day 1 Post LAIV
Description: No of participants with viral shedding on day 1 following LAIV vaccination
Time Frame: Assessed on day 1 post LAIV
Measure: Count of Participants; unit: Participants
Arm/Group | All Children
Number analyzed (Participants) | 12
Participants | 3

2. Primary Outcome: Type-specific Vaccine Virus Shedding in 2018/19 - Day 2 Post LAIV
Description: No of participants with viral shedding on day 2 following LAIV vaccination
Time Frame: Assessed on day 2 post LAIV
Measure: Count of Participants; unit: Participants
Arm/Group | All Children
Number analyzed (Participants) | 12
Participants | 3

3. Primary Outcome: Type-specific Vaccine Virus Shedding in 2018/19 - Day 3 Post LAIV
Description: No of participants with viral shedding on day 3 following LAIV vaccination
Time Frame: Assessed on day 3 post LAIV
Measure: Count of Participants; unit: Participants
Arm/Group | All Children
Number analyzed (Participants) | 12
Participants | 1

4. Primary Outcome: Type-specific Vaccine Virus Shedding in 2018/19 - Day 4 Post LAIV
Description: No of participants with viral shedding on day 4 following LAIV vaccination
Time Frame: Assessed on day 4 post LAIV
Measure: Count of Participants; unit: Participants
Arm/Group | All Children
Number analyzed (Participants) | 12
Participants | 3

5. Primary Outcome: Type-specific Vaccine Virus Shedding in 2018/19 - Day 5 Post LAIV
Description: No of participants with viral shedding on day 5 following LAIV vaccination
Time Frame: Assessed on day 5 post LAIV
Measure: Count of Participants; unit: Participants
Arm/Group | All Children
Number analyzed (Participants) | 12
Participants | 3

6. Primary Outcome: Type-specific Vaccine Virus Shedding in 2018/19 - Day 6 Post LAIV
Description: No of participants with viral shedding on day 6 following LAIV vaccination
Time Frame: Assessed on day 6 post LAIV
Measure: Count of Participants; unit: Participants
Arm/Group | All Children
Number analyzed (Participants) | 12
Participants | 3

7. Primary Outcome: Type-specific Vaccine Virus Shedding in 2018/19 - Day 7 Post LAIV
Description: No of participants with viral shedding on day 7 following LAIV vaccination
Time Frame: Assessed on day 7 post LAIV
Measure: Count of Participants; unit: Participants
Arm/Group | All Children
Number analyzed (Participants) | 12
Participants | 2

8. Primary Outcome: Type-specific Vaccine Virus Shedding in 2018/19 - Day 8 Post LAIV
Description: No of participants with viral shedding on day 8 following LAIV vaccination
Time Frame: Assessed on day 8 post LAIV
Measure: Count of Participants; unit: Participants
Arm/Group | All Children
Number analyzed (Participants) | 12
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse events up to Day 8 after LAIV. SAEs up to Day 28.
Arm/Group | All Children
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/47/NCT03735147/Prot_SAP_000.pdf